CLINICAL TRIAL: NCT05588219
Title: Tislelizumab Combined With Concurrent Chemoradiotherapy for Locally Advanced Cervical Cancer: a Prospective, Single-arm, Single-center, Phase II Clinical Study
Brief Title: Tislelizumab Combined With Concurrent Chemoradiotherapy for Locally Advanced Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yong Zhang,MD (Other)
Responsible Party: Sponsor-Investigator, Yong Zhang,MD, First Affiliated Hospital of Guangxi Medical University, First Affiliated Hospital of Guangxi Medical University
Organization: First Affiliated Hospital of Guangxi Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-K046-01
Record Dates: First submitted 2022-10-18; First posted 2022-10-20 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Cervical cancer; Tislelizumab; Concurrent chemoradiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — tislelizumab; Immune Checkpoint Inhibitors; Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): The therapeutic schedule of the experimental arm: External irradiation 45~50Gy/25f+ Brachytherapy 28~30Gy/4~5f; Chemotherapy: DDP 40mg/m2/W, synchronous with radiotherapy, complete at least 4 cycles; Tislelizumab injection[10ml:100mg]: 200mg/3W for 1 year or disease progression or intolerable toxicity, whichever occurs first.
  Interventions: Drug: Tislelizumab; Drug: DDP synchronous with radiotherapy

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab injection[10ml:100mg] will be used beginning with radiotherapy: 200mg/3W for 1 year or disease progression or intolerable toxicity, whichever occurs first.
  Other Names: Immune checkpoint inhibitors
Drug: DDP synchronous with radiotherapy — DDP 40mg/m2/W, synchronous with radiotherapy, complete at least 4 cycles.
  Other Names: Cisplatin

SUMMARY:
This study aims to evaluate the efficacy and safety of Tislelizumab combined with concurrent chemoradiotherapy in the treatment of cervical cancer patients with cervical mass > 4cm and regional lymph node metastasis, paracervical invasion and regional lymph node metastasis, stage IIIA, stage IIIB, and stage IVA. To provide a clinical reference for finding a safe and effective individualized treatment plan to improve the survival prognosis of locally advanced cervical cancer patients.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center phase II clinical study. The objective is to evaluate the efficacy and safety of Tislelizumab combined with concurrent chemoradiotherapy in the treatment of locally advanced cervical cancer. This study was independently completed by our center. Cervical cancer patients with cervical mass > 4cm with regional lymph node metastasis, paracervical invasion with regional lymph node metastasis, stage IIIA, stage IIIB and stage IVA in FIGO stage 2018 were selected as subjects, and 30 patients were planned to be enrolled. External irradiation 45~50Gy/25f+ Brachytherapy 28~30Gy/4~5f; Chemotherapy: DDP 40mg/m2/W, synchronous with radiotherapy, complete at least 4 cycles; Tislelizumab: 200mg/3W for 1 year or disease progression or intolerable toxicity, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years.
2. The pathological types of cervical cancer confirmed by histopathology were squamous cell carcinoma, adenocarcinoma and adenosquamous cell carcinoma.
3. In FIGO stage 2018, cervical mass > 4cm with regional lymph node metastasis, paracervical invasion with regional lymph node metastasis, stage IIIA, stage IIIB, and stage IVA.
4. Having at least one measurable lesion according to RECIST 1.1.
5. ECOG score 0-1.
6. Expected survival time ≥6 months.
7. Major organ function is normal, that is, meeting the following criteria: blood routine: HB≥90g/L, ANC≥1.5×109/L, PLT≥80×109/L; Biochemical examination of ALB≥30g/L, TBIL≤1.5 ULN, ALT and AST≤2.5 ULN, plasma Cr≤1.5 ULN or creatinine clearance ≥60 ml/min.
8. Menopausal women, or women of childbearing age who meet all the following conditions: non-lactation, not pregnant, and can take adequate contraceptive measures during the study treatment.
9. Subjects volunteered to join the study, signed the informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Patients have had or currently have other malignant tumors within 5 years.
2. Patients allergic or sensitive to any drug in the study protocol.
3. Patients innate or acquired immune deficiency (e.g. HIV infection).
4. The presence of any active, known or suspected autoimmune disease (such as, but not limited to, interstitial pneumonia, uveitis, enteritis, hepatitis, arthritis, nephritis, hypophysitis, hyperthyroidism, hypothyroidism, etc.); The subject had vitiligo. Subjects with asthma require bronchodilators for medical intervention.
5. The presence of active infections requiring systemic treatment.
6. The subject has previously received other PD-1 or PD-L1, or CTLA-4 antibody therapy, or other drug therapy targeting immunoregulatory receptor preparations.
7. Unrelieved toxic effects above CTCAE grade 1 due to any previous treatment, excluding alopecia.
8. Patients with a history of myocardial infarction or stroke, unstable angina pectoris, decompensated heart failure or deep vein thrombosis.
9. Patients with long-term untreated wounds or fractures, major surgical operations or severe traumatic injuries, fractures or ulcers within 4 weeks.
10. Pregnant or lactating women.
11. Patients with liver and kidney dysfunction.
12. Patients with a history of abuse of psychotropic drugs and unable to abstain or patients with mental disorders.
13. Patients who have participated in clinical trials of other drugs within 4 weeks.
14. Patients with concomitant diseases that, in the judgment of the investigator, seriously endanger the patient's safety or affect the patient's completion of the study.
15. The investigator judged that participation in this study was not conducive to the maximum benefit of the subjects.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor regression ratio | 2 weeks
  The tumor regression ratio after external irradiation, MRI/CT will be used for evaluating the carcinoma status.

SECONDARY OUTCOMES:
Overall Response Rate | 3 months, 6 moths
  The overall response rate or tumor after radiotherapy and chemotherapy, and MRI/CT will be used for evaluating the carcinoma status.
Overall Survival | 1 years, 3 years
  OS was calculated from the date of entry into the study to the date of death or the last follow-up visit.
Progression Free Survival | 1 years, 3 years
  PFS was calculated from the date of entry into the study to the date of first physical or radio-graphic evidence of disease progression, death or the last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Songqing He, PhD, Study Chair — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No